CLINICAL TRIAL: NCT05035147
Title: Non-inferiority Study of Albumin-bound Paclitaxel Combined With Gemcitabine for Three Weeks Versus Four Weeks for First-line Inoperable Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Albumin-bound Paclitaxel Combined With Gemcitabine First-line Inoperable Pancreatic Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJGI-003
Record Dates: First submitted 2021-08-16; First posted 2021-09-05 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose strength: albumin-bound paclitaxel + gemcitabine (Experimental): albumin-bound paclitaxel 125mg/m2+ gemcitabine1000mg/m2:day1,8 q3w
  Interventions: Drug: albumin-bound paclitaxel
- High dose strength: albumin-bound paclitaxel + gemcitabine (Active Comparator): albumin-bound paclitaxel 125mg/m2+ gemcitabine1000mg/m2:day1,8,15 q4w
  Interventions: Drug: albumin-bound paclitaxel

INTERVENTIONS:
Drug: albumin-bound paclitaxel — Experimental:Albumin-bound paclitaxel combined with gemcitabine was administered on the first and eighth day, a cycle of three weeks Active Comparator: Albumin-bound paclitaxel combined with gemcitabine was administered on the first, eighth, and fifteenth days, with a four-week cycle
  Other Names: gemcitabine

SUMMARY:
This study aims to further observe and evaluate whether the three-week administration of albumin-bound paclitaxel combined with gemcitabine is equivalent to the four-week administration in the treatment of inoperable locally advanced or metastatic pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer is a common clinical malignant tumor of the digestive system, and its incidence is gradually increasing worldwide.The prognosis is poor and the mortality rate is high, accounting for about 7% of cancer deaths.Albumin-bound paclitaxel is a good first-line treatment for pancreatic cancer. It has the advantages of high dose, high tumor tissue distribution, high efficacy, and low toxicity.It is hoped that the low-dose intensity can achieve the same clinical efficacy as the high-dose intensity, which provides strong evidence for the clinical choice of low-dose intensity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, no gender limit;
2. Inoperable locally advanced or metastatic pancreatic cancer patients (except islet cell carcinoma) diagnosed by pathology or histology;
3. The patient has not undergone standard systemic treatment in the past, or more than half a year after the end of postoperative treatment.For those who have undergone major surgery or radiotherapy, the interval must be more than 4 weeks and their metastases have not received any local treatment including radiotherapy, chemotherapy, surgical treatment, etc.;
4. At least one measurable lesion (CT scan of tumor lesions with long diameter ≥ 10 mm, CT scan of lymph node lesions with short diameter ≥ 15 mm, and scan thickness not greater than 6 mm);
5. The main organs are functioning normally, that is, they meet the following standards:Routine blood examination: Hb≥90g/L (no blood transfusion within 14 days);ANC ≥1.5×109/L;PLT ≥100×109/L;Biochemical examination: ALB≥29 g/L (without ALB in 14 days), TBIL <1.5 times the upper limit of normal (ULN);ALT and AST≤3ULN, accompanied by liver metastasis, then ALT and AST<5×ULN;Cr ≤1.5×ULN or creatinine clearance rate ≥60ml/min;
6. The subject voluntarily joined the study and signed an informed consent form, with good compliance and cooperation with follow-up

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients suffering from other malignant tumors in the past or at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
3. Those who have been confirmed to be allergic to the test drug albumin-bound paclitaxel and gemcitabine or its excipients.
4. The patient has clinically significant ascites;
5. Those who have experienced arterial/venous thrombosis within six months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
6. Patients with active hepatitis B or C;
7. Doctors think it is not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | through study completion, an average of 5year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | through study completion, an average of 5year
  The percentage of confirmed complete remission, partial remission and stable disease among patients with evaluable efficacy
Objective response rate(ORR) | through study completion, an average of 5year
  The proportion of patients whose tumors have shrunk to a certain level and maintained for a certain period of time, including CR and PR cases.The solid tumor response assessment standard (RECIST 1.1 standard) was used to assess the objective tumor response.The subject must have measurable tumor lesions at baseline.According to the RECIST 1.1 standard, the efficacy evaluation criteria are divided into complete remission (CR), partial remission (PR), stable (SD), and progress (PD)
Overall survival(OS) | through study completion, an average of 5year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ji zhi, professor, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Rui Liu, Tianjin, Tianjin Municipality, China